CLINICAL TRIAL: NCT06492226
Title: A Single-center, Single-dose, Double-blind, Randomized, Three-period, Three-treatment, Six-sequence, Crossover Study to Demonstrate Pharmacokinetic and Pharmacodynamic Similarity Between NKF-INS(A), US-NovoLog®, and EU-NovoRapid® Using the Euglycemic Clamp Technique in Healthy Male Adult Volunteers
Brief Title: Study to Demonstrate Pharmacokinetic and Pharmacodynamic Similarity Between NKF-INS(A), US-NovoLog®, and EU-NovoRapid®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NKF-INS(A)-101
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- NKF-INS(A) (Experimental): Single subcutaneous dose administration over three treatment periods
  Interventions: Drug: NKF-INS(A)
- EU-NovoRapid® (Active Comparator): Single subcutaneous dose administration over three treatment periods
  Interventions: Drug: EU-NovoRapid®
- US-NovoLog® (Active Comparator): Single subcutaneous dose administration over three treatment periods
  Interventions: Drug: US-NovoLog®

INTERVENTIONS:
Drug: NKF-INS(A) — Single subcutaneous dose of 0.3 U/kg administration over three treatment periods
  Arms: NKF-INS(A)
Drug: EU-NovoRapid® — Single subcutaneous dose of 0.3 U/kg administration over three treatment periods
  Arms: EU-NovoRapid®
Drug: US-NovoLog® — Single subcutaneous dose of 0.3 U/kg administration over three treatment periods
  Arms: US-NovoLog®

SUMMARY:
Single-dose, double-blind, randomized, three-period, three-treatment, six-sequence, crossover study to demonstrate pharmacokinetic and pharmacodynamic similarity between NKF-INS(A), US-NovoLog®, and EU-NovoRapid®

DETAILED DESCRIPTION:
A single-center, single-dose, double-blind, randomized, three-period, three-treatment, six-sequence, crossover study to demonstrate pharmacokinetic and pharmacodynamic similarity between NKF-INS(A), US-NovoLog®, and EU-NovoRapid® using the euglycemic clamp technique in healthy male adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial-related activities. Trial-related activities are any procedures that would not have been done during normal management of the participant
2. Healthy male participants
3. Age between 18 and 50 years, both inclusive
4. Body Mass Index between 18.5 and 29.0 kg/m2, both inclusive
5. Body weight ≥ 50 kg
6. Fasting plasma glucose concentration ≤ 5.5 mmol/L at screening
7. Considered generally healthy upon completion of medical history, physical examination, vital signs, electrocardiogram (ECG), and analysis of laboratory safety variables, as judged by the Investigator
8. Willing and able to comply with scheduled visits, treatment plan, clinical laboratory tests, and other study procedures including lifestyle considerations.
9. Participants must agree to use condoms during sexual intercourse. Additionally, female partners of male participants should use highly effective contraception. All contraceptive measures apply from screening until 90 days after study
10. Have competence in speaking, writing, and comprehending the local language(s) where the study is conducted.

Exclusion Criteria:

1. Positive for human insulin antibodies at Screening
2. Are currently enrolled in or have discontinued within 3 months or 5 half-lives (whichever is longer) of any investigational drug or device or are concurrently enrolled in any other type of medical research study and judged not to be scientifically or medically compatible with this study.
3. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.
4. History of diabetes mellitus; episodes of hypoglycemia in the anamnesis; any history of insulin use for treatment purposes.
5. Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin.
6. Have clinically relevant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study drug; or of interfering with the interpretation of data.
7. Increased risk of thrombosis, e.g., individuals with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.
8. Clinically significant abnormal ECG at screening.
9. Glycemia level ≥140.4 mg/dL 2 hours after the glucose load.
10. Show evidence of significant active neuropsychiatric disease.
11. Positive urine drug test at screening and/or evidence of current use of known drugs of abuse or have a history of use within the past year.
12. Show evidence of an acute infection with fever or infectious disease at the time of enrollment.
13. Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening.
14. Have positive test results for hepatitis B surface antigen (HBsAg), immunoglobulin M (IgM) antibody to hepatitis B core antigen (anti-HBc), or hepatitis C virus (HCV) antibodies at screening.
15. Intend to use over-the-counter medication within 7 days or prescription medication within 14 days prior to dosing (apart from vitamin/mineral supplements, occasional paracetamol, thyroid replacement).
16. Have donated blood or had a blood loss of 450 mL 3 months prior to study enrollment.
17. Have an average weekly alcohol intake that exceeds 21 units per week or is unwilling to stop alcohol consumption from 48 hours prior to each dosing until being discharged from the CRU.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Xentria Investigative Site, Bloemfontein, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NKF-INS(A), EU-NovoRapid, US-NovoLog: Participants first received NKF-INS(A) on Day 1 of Treatment Period 1. After a washout period of 3-14 calendar days, they then received EU-NovoRapid on Day 1 of Treatment Period 2. After an additional washout period of 5-21 calendar days, they then received US-NovoLog on Day 1 of Treatment Period 3.
- NKF-INS(A), US-NovoLog, EU-NovoRapid: Participants first received NKF-INS(A) on Day 1 of Treatment Period 1. After a washout period of 3-14 calendar days, they then received US-NovoLog on Day 1 of Treatment Period 2. After an additional washout period of 5-21 calendar days, they then received EU-NovoRapid on Day 1 of Treatment Period 3.
- EU-NovoRapid, NKF-INS(A), US-NovoLog: Participants first received EU-NovoRapid on Day 1 of Treatment Period 1. After a washout period of 3-14 calendar days, they then received NKF-INS(A) on Day 1 of Treatment Period 2. After an additional washout period of 5-21 calendar days, they then received US-NovoLog on Day 1 of Treatment Period 3.
- EU-NovoRapid, US-NovoLog, NKF-INS(A): Participants first received EU-NovoRapid on Day 1 of Treatment Period 1. After a washout period of 3-14 calendar days, they then received US-NovoLog on Day 1 of Treatment Period 2. After an additional washout period of 5-21 calendar days, they then received NKF-INS(A) on Day 1 of Treatment Period 3.
- US-NovoLog, NKF-INS(A), EU-NovoRapid: Participants first received US-NovoLog on Day 1 of Treatment Period 1. After a washout period of 3-14 calendar days, they then received NKF-INS(A) on Day 1 of Treatment Period 2. After an additional washout period of 5-21 calendar days, they then received EU-NovoRapid on Day 1 of Treatment Period 3.
- US-NovoLog, EU-NovoRapid, NKF-INS(A): Participants first received US-NovoLog on Day 1 of Treatment Period 1. After a washout period of 3-14 calendar days, they then received EU-NovoRapid on Day 1 of Treatment Period 2. After an additional washout period of 5-21 calendar days, they then received NKF-INS(A) on Day 1 of Treatment Period 3.
Period: Overall Study
Arm/Group | NKF-INS(A), EU-NovoRapid, US-NovoLog | NKF-INS(A), US-NovoLog, EU-NovoRapid | EU-NovoRapid, NKF-INS(A), US-NovoLog | EU-NovoRapid, US-NovoLog, NKF-INS(A) | US-NovoLog, NKF-INS(A), EU-NovoRapid | US-NovoLog, EU-NovoRapid, NKF-INS(A)
Started | 9 | 9 | 9 | 9 | 9 | 9
Completed | 8 | 9 | 8 | 9 | 9 | 9
Not Completed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NKF-INS(A), US-NovoLog-EU, NovoRapid: Participants first received NKF-INS(A) on Day 1 of Treatment Period 1. After a washout period of 3-14 calendar days, they then received US-NovoLog on Day 1 of Treatment Period 2. After an additional washout period of 5-21 calendar days, they then received EU-NovoRapid on Day 1 of Treatment Period 3.
- Total: Total of all reporting groups
Arm/Group | NKF-INS(A), EU-NovoRapid, US-NovoLog | NKF-INS(A), US-NovoLog-EU, NovoRapid | EU-NovoRapid, NKF-INS(A), US-NovoLog | EU-NovoRapid, US-NovoLog, NKF-INS(A) | US-NovoLog, NKF-INS(A), EU-NovoRapid | US-NovoLog, EU-NovoRapid, NKF-INS(A) | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 54
Age, Customized [Mean (Standard Deviation); unit: years] | 36.3 (6.2) | 30.2 (6.3) | 34.2 (9.8) | 32.1 (5.7) | 30.4 (8.4) | 35.1 (7.8) | 33.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 9 | 9 | 9 | 9 | 9 | 9 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 8 | 9 | 6 | 9 | 7 | 6 | 45
  Other | 0 | 0 | 2 | 0 | 0 | 1 | 3
  White | 1 | 0 | 1 | 0 | 2 | 2 | 6
  Not Hispanic or Latino | 9 | 9 | 9 | 9 | 9 | 9 | 54
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 25.1 (2.9) | 24.7 (2.1) | 24.3 (2.7) | 23.9 (2.1) | 24.7 (2.0) | 23.7 (2.7) | 24.4 (2.4)
Height (cm) [Mean (Standard Deviation); unit: cm] | 171.6 (8.9) | 172.2 (7.9) | 173.9 (7.4) | 172.6 (3.9) | 172.4 (7.3) | 171.0 (9.4) | 172.3 (7.4)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 73.9 (8.8) | 73.5 (10.6) | 73.4 (10.2) | 71.4 (7.1) | 73.6 (7.7) | 69.0 (6.9) | 72.5 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Aspart Concentration-time Curve From 0 to 12 Hours Area Under the Insulin Aspart Concentration-Time Curve (AUC0-t).
Description: Compared the Pharmacokinetics (PK) of NKF-INS(A) to United States (US)-approved and European Union (EU)-authorized insulin aspart demonstrating PK similarity for insulin aspart.
Time Frame: Day 1 for 12 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/ml
Groups:
- EU-NovoRapid®; US-NovoLog®; NKF-INS(A): Participants received a single subcutaneous dose of 0.3 IU/kg in either Treatment Period 1, Treatment Period 2, or Treatment Period 3
Arm/Group | EU-NovoRapid® | US-NovoLog® | NKF-INS(A)
Number analyzed (Participants) | 52 | 52 | 52
min*ng/ml | 894.971 (18.426) | 899.163 (18.711) | 904.131 (17.174)
Statistical Analysis 1: Comparison: EU-NovoRapid® vs NKF-INS(A); Test type: Equivalence — Biosimilarity of the test and reference products was assessed on the basis of the 95% CIs for estimates of the geometric mean ratios between the primary PK parameters of the test and reference products in relation to the conventional bioequivalence range of 80% to 125%; Geometric Mean Ratio = 101.024, 95% CI 2-sided [98.754 to 103.346]
Statistical Analysis 2: Comparison: US-NovoLog® vs NKF-INS(A); Test type: Equivalence — Biosimilarity of the test and reference products was assessed on the basis of the 90% CIs for estimates of the geometric mean ratios between the primary PK parameters of the test and reference products in relation to the conventional bioequivalence range of 80% to 125%; Geometric Mean Ratio = 100.682, 90% CI 2-sided [98.567 to 102.843]

2. Primary Outcome: Maximum Observed Insulin Aspart Concentration Maximum Observed Insulin Aspart Concentration (Cmax)
Description: Compared the Pharmacokinetic (PK) of NKF-INS(A) to United States (US)-approved and European Union (EU)-authorized insulin aspart demonstrating PK similarity for insulin aspart.
Time Frame: Day 1 for 12 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | EU-NovoRapid® | US-NovoLog® | NKF-INS(A)
Number analyzed (Participants) | 52 | 52 | 52
ng/ml | 1.754 (16.331) | 1.754 (17.492) | 1.805 (15.255)
Statistical Analysis 1: Comparison: EU-NovoRapid® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 104.931, 95% CI 2-sided [99.630 to 110.514]
Statistical Analysis 2: Comparison: US-NovoLog® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Geometric Mean Ratio = 105.000, 90% CI 2-sided [100.827 to 109.345]

3. Primary Outcome: Area Under the GIR-time Curve From 0 to 12 Hours (AUCGIR0-t).
Description: Compared the Pharmacodynamic (PD) of NKF-INS(A) to United States (US)-approved and European Union (EU)-authorized insulin aspart injection by examining Glucose Infusion Rate (GIR) profiles after a single Subcutaneous (SC) dose.
Time Frame: Day 1 for 12 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*mg/min
Arm/Group | EU-NovoRapid® | US-NovoLog® | NKF-INS(A)
Number analyzed (Participants) | 52 | 52 | 52
min*mg/min | 166278.835 (25.467) | 167245.347 (26.287) | 171020.184 (26.779)
Statistical Analysis 1: Comparison: EU-NovoRapid® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 102.851, 95% CI 2-sided [96.749 to 109.339]
Statistical Analysis 2: Comparison: US-NovoLog® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Geometric Mean Ratio = 102.006, 90% CI 2-sided [97.308 to 106.930]

4. Primary Outcome: Maximum GIR (GIRmax) of Glucose
Description: as for outcome 3
Time Frame: Day 1 for 12 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/min
Arm/Group | EU-NovoRapid® | US-NovoLog® | NKF-INS(A)
Number analyzed (Participants) | 52 | 52 | 52
mg/min | 604.789 (26.670) | 619.459 (29.184) | 608.934 (26.825)
Statistical Analysis 1: Comparison: EU-NovoRapid® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 100.685, 95% CI 2-sided [94.956 to 106.760]
Statistical Analysis 2: Comparison: US-NovoLog® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Geometric Mean Ratio = 97.980, 90% CI 2-sided [92.554 to 103.723]

5. Secondary Outcome: PK Parameters for Serum Insulin Aspart Concentrations: Area Under the Insulin Aspart Concentration-Time Curve (AUC0)-4h, AUC0-6h, AUC0-12h, AUC0-∞
Description: Evaluated additional Pharmacokinetic (PK) parameters of NKF-INS(A) compared to United Stated (US)-approved and European Union (EU)-authorized insulin aspart.
Time Frame: Day 1 for 12 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | EU-NovoRapid® | US-NovoLog® | NKF-INS(A)
Number analyzed (Participants) | 52 | 52 | 52
min*ng/mL
  Area Under the Insulin Aspart Concentration-Time Curve (AUC0 -4h) | 828.375 (19.345) | 834.396 (20.308) | 845.061 (17.616)
  Area Under the Insulin Aspart Concentration-Time Curve (AUC0 -6h) | 891.162 (18.308) | 899.163 (18.711) | 899.437 (17.172)
  Area Under the Insulin Aspart Concentration-Time Curve AUC0-12h | 894.971 (18.426) | 899.163 (18.711) | 904.131 (17.174)
  Area Under the Insulin Aspart Concentration-Time Curve AUC0-∞ | 965.874 (19.327) | 988.791 (19.146) | 959.327 (17.480)
Statistical Analysis 1: Comparison: EU-NovoRapid® vs NKF-INS(A); PK parameters for serum insulin aspart concentrations: Area Under the Insulin Aspart Concentration-Time Curve (AUC0)-4h; Test type: Equivalence — Biosimilarity of the test and reference products was assessed on the basis of the 95% CIs for estimates of the geometric mean ratios between the PK parameters of the test and reference products in relation to the conventional bioequivalence range of 80% to 125%; Geometric Mean Ratio = 102.014, 95% CI 2-sided [99.090 to 105.025]
Statistical Analysis 2: Comparison: US-NovoLog® vs NKF-INS(A); PK parameters for serum insulin aspart concentrations: Area Under the Insulin Aspart Concentration-Time Curve (AUC0)-4h; Test type: Equivalence — Biosimilarity of the test and reference products was assessed on the basis of the 90% CIs for estimates of the geometric mean ratios between the PK parameters of the test and reference products in relation to the conventional bioequivalence range of 80% to 125%; Geometric Mean Ratio = 101.419, 90% CI 2-sided [99.062 to 103.833]
Statistical Analysis 3: Comparison: EU-NovoRapid® vs NKF-INS(A); PK parameters for serum insulin aspart concentrations: Area Under the Insulin Aspart Concentration-Time Curve AUC0-6h; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Geometric Mean Ratio = 100.929, 95% CI 2-sided [98.393 to 103.529]
Statistical Analysis 4: Comparison: US-NovoLog® vs NKF-INS(A); PK parameters for serum insulin aspart concentrations: Area Under the Insulin Aspart Concentration-Time Curve AUC0-6h; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric Mean Ratio = 100.127, 90% CI 2-sided [98.080 to 102.217]
Statistical Analysis 5: Comparison: EU-NovoRapid® vs NKF-INS(A); PK parameters for serum insulin aspart concentrations: Area Under the Insulin Aspart Concentration-Time Curve AUC0-12h; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Geometric Mean Ratio = 101.024, 95% CI 2-sided [98.754 to 103.346]
Statistical Analysis 6: Comparison: US-NovoLog® vs NKF-INS(A); PK parameters for serum insulin aspart concentrations: Area Under the Insulin Aspart Concentration-Time Curve AUC0-12h; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric Mean Ratio = 100.682, 90% CI 2-sided [98.567 to 102.843]
Statistical Analysis 7: Comparison: EU-NovoRapid® vs NKF-INS(A); PK parameters for serum insulin aspart concentrations: Area Under the Insulin Aspart Concentration-Time Curve AUC0-∞; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Geometric Mean Ratio = 98.881, 95% CI 2-sided [96.400 to 101.426]
Statistical Analysis 8: Comparison: US-NovoLog® vs NKF-INS(A); PK parameters for serum insulin aspart concentrations: Area Under the Insulin Aspart Concentration-Time Curve AUC0-∞; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric Mean Ratio = 97.023, 90% CI 2-sided [94.863 to 99.232]

6. Secondary Outcome: Time to Half-maximum Before Maximum Observed Insulin Aspart Concentration Time to Half-Maximum Before Maximum Observed Insulin Aspart Concentration (t50%-Early)
Description: Evaluated Additional Pharmacokinetic (PK) Parameters of NKF-INS(A) Compared to United States (US)-Approved and European (EU)-Authorized Insulin Aspart.
Time Frame: Day 1 for 12 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: minutes
Arm/Group | EU-NovoRapid® | US-NovoLog® | NKF-INS(A)
Number analyzed (Participants) | 52 | 52 | 52
minutes | 24.515 (22.919) | 26.597 (25.395) | 21.980 (27.890)
Statistical Analysis 1: Comparison: EU-NovoRapid® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Geometric Mean Ratio = 89.656, 95% CI 2-sided [84.557 to 95.064]
Statistical Analysis 2: Comparison: US-NovoLog® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric Mean Ratio = 82.086, 90% CI 2-sided [76.699 to 87.851]

7. Secondary Outcome: Time to Half-maximum After Maximum Observed Insulin Aspart Concentration Time to Half-Maximum After Maximum Observed Insulin Aspart Concentration (t50%-Late)
Description: as for outcome 5
Time Frame: Day 1 for 12 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: minutes
Arm/Group | EU-NovoRapid® | US-NovoLog® | NKF-INS(A)
Number analyzed (Participants) | 52 | 52 | 52
minutes | 169.891 (30.545) | 177.331 (29.442) | 161.226 (27.896)
Statistical Analysis 1: Comparison: EU-NovoRapid® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Geometric Mean Ratio = 94.900, 95% CI 2-sided [89.997 to 100.070]
Statistical Analysis 2: Comparison: US-NovoLog® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric Mean Ratio = 90.601, 90% CI 2-sided [86.356 to 95.054]

8. Secondary Outcome: The Terminal Elimination Half-life (t1/2)
Description: as for outcome 5
Time Frame: Day 1 for 12 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: minutes
Arm/Group | EU-NovoRapid® | US-NovoLog® | NKF-INS(A)
Number analyzed (Participants) | 46 | 46 | 46
minutes | 55.742 (38.083) | 58.096 (47.795) | 53.348 (33.361)
Statistical Analysis 1: Comparison: EU-NovoRapid® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Geometric Mean Ratio = 95.232, 95% CI 2-sided [88.411 to 102.580]
Statistical Analysis 2: Comparison: US-NovoLog® vs NKF-INS(A); Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric Mean Ratio = 91.300, 90% CI 2-sided [83.291 to 100.079]

9. Secondary Outcome: PK Parameters for Serum Insulin Aspart Concentrations: Area Under the Insulin Aspart Concentration-Time Curve to Maximum Insulin Aspart Concentration (Tmax)
Description: as for outcome 5
Time Frame: Day 1 for 12 Hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: minutes
Arm/Group | EU-NovoRapid® | US-NovoLog® | NKF-INS(A)
Number analyzed (Participants) | 52 | 52 | 52
minutes | 64.411 (37.344) | 69.888 (37.380) | 53.904 (34.668)
Statistical Analysis 1: Comparison: EU-NovoRapid® vs NKF-INS(A); Test type: Equivalence — Biosimilarity of the test and reference products was assessed on the basis of the 95% CIs for estimates of the geometric mean ratios between the PK parameters of the test and reference products; Geometric Mean Ratio = 83.687, 95% CI 2-sided [76.783 to 91.213]
Statistical Analysis 2: Comparison: US-NovoLog® vs NKF-INS(A); Test type: Equivalence — Biosimilarity of the test and reference products was assessed on the basis of the 90% CIs for estimates of the geometric mean ratios between the PK parameters of the test and reference products; Geometric Mean Ratio = 76.497, 90% CI 2-sided [69.750 to 83.897]

10. Secondary Outcome: PK Parameters for Serum Insulin Aspart Concentrations: Area Under the Insulin Aspart Concentration-Time Curve AUC6-12h
Description: as for outcome 5
Time Frame: Day 1 for 12 Hours
Population: The Pharmacokinetic Parameter for the 6-12 hour interval [(6-Inf(hrs): AUC0-t(min*ng/ml)] only contains two participants due to only two participants recording an Aspart concentration above the lower limit of quantification beyond 6 hours. All other participants did not record a quantifiable concentration between 6 and 12 hours. Therefore, this PK parameter was not included in the bioequivilance assessment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/ml
Arm/Group | EU-NovoRapid® | NKF-INS(A)
Number analyzed (Participants) | 1 | 1
min*ng/ml | 36.36 (NA) — Only 2 participants recorded an Aspart concentration above the lower limit of quantification beyond 6 hours. The measure of dispersion/precision is not available as standard deviation is not calculable for 1 participant. All other participants did not record a quantifiable concentration between 6 and 12 hours. Therefore, this PK parameter was not included in the bioequivilance assessment. | 30.360 (NA) — Only 2 participants recorded an Aspart concentration above the lower limit of quantification beyond 6 hours. The measure of dispersion/precision is not available as standard deviation is not calculable for 1 participant. All other participants did not record a quantifiable concentration between 6 and 12 hours. Therefore, this PK parameter was not included in the bioequivilance assessment.

ADVERSE EVENTS:
Time Frame: Beginning of study treatment (Day 1) until the End of Study Visit (within 2-11 days of last administration of study drug). Adverse event (AE) assessments (including injection site reactions), clinical laboratory investigations (hematology, clinical chemistry [including glucose], coagulation, and urinalysis), vital signs, physical examinations, 12-lead electrocardiogram (ECG), prior and concomitant medication assessments
Description: Three insulin products (NKF-INS(A), EU-NovoRapid, and US-NovoLog) were administered over three treatment periods. Participants were randomized to one of six treatment sequences in a 1:1:1:1:1:1 ratio, receiving a single SC dose of 0.3 international units (IU)/kg administration of one of the three study drugs on each dosing day. All enrolled participants who completed the study received each of the 3 treatments over their 3 treatment periods
Arm/Group | NKF-INS(A) | EU-NovoRapid® | US-NovoLog®
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 8/53 | 6/53 | 4/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NKF-INS(A) (N=53) | EU-NovoRapid® (N=53) | US-NovoLog® (N=52)
Headache (Nervous system disorders) | 3 | 1 | 3
Thrombophlebitis (Vascular disorders) | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Infusion site pain (General disorders) | 1 | 0 | 0
Shoulder girdle pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT06492226/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT06492226/SAP_001.pdf